CLINICAL TRIAL: NCT06687798
Title: Validation of a Questionnaire to Evaluate the Home Cooking Skills of Nutrition Professionals and the General Population (HCSQ-ITA)
Brief Title: Validation of a Questionnaire to Evaluate the Home Cooking Skills of Nutrition Professionals and the General Population
Acronym: HCSQ-ITA
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pavia (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: 65372/2023
Record Dates: First submitted 2024-02-20; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-02

CONDITIONS: Cooking
Keywords: cooking; Health Personnel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to validate the questionnaire HCSQ-ITA in nutrition students and professionals (dieticians, biologists-nutritionists, medical specialists in food science, and experts in gastronomic techniques) or the general population.

The main question it aims to answer is:

- Is the questionnaire to evaluate the cooking skills of nutrition professionals valid? Participants will answer an electronic form questionnaire (HCSQ-ITA) and evaluate its clarity and pertinence.

DETAILED DESCRIPTION:
Unbalanced food choices are a major determinant of the global disease burden, with one in five deaths worldwide attributable to an inadequate diet. Food patterns characterized by reduced consumption of whole grains, fruits, vegetables, dried fruit, and legumes, along with excessive sodium, red or processed meats, and sugary foods, are associated with a high risk of developing chronic non-communicable diseases (NCDs), such as cancer, cardiovascular diseases, and diabetes. High adherence to healthy dietary patterns, such as the Mediterranean Diet, is associated with a lower risk of diabetes, cardiovascular disease, cancer, and cognitive decline. However, global populations are gradually reducing their adherence to this dietary pattern, preferring diets rich in saturated fats and animal-derived protein. This phenomenon, known as the nutritional transition, is associated with a concomitant culinary transition, a progressive change in cooking skills required for home-made meals. Improving culinary skills can have a positive impact on food choices and the quality of the diet. Nutrition professionals can play a crucial role in promoting food and nutrition education initiatives and actions, providing practical experiences and suggestions to help change eating habits. The study aims to validate the Primary Health Care Home Cooking Skills Scale, already validated in Brazil; tool for a representative sample of the general population and nutrition professionals in Italy.

The process of validation will include several stages: (1) the validated Brazilian questionnaire will be translated and adapted to the content. After this, the (2) validation of the content will follow Delphi's technique, and then (2) analysis of the validity and (3) reliability of the construction, through the factor analysis.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years and ≤ 65 years,
* all genres
* signature of informed consent
* nutrition students and professionals (dieticians, biologists-nutritionists, medical specialists in food science and experts in gastronomic techniques)
* general population (non-nutrition professionals)

Exclusion Criteria:

* Serious physical and psychiatric illnesses
* Disorders requiring treatment with atypical antipsychotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: -Healthy adults, all genres, nutrition students and professionals (dieticians, biologists-nutritionists, medical specialists in food science and experts in gastronomic techniques)
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Home cooking skills | 6 months
  The final score will classify the sample according to the cooking skills with the "Home cooking skills questionnaire - Italian version" (HCSQ-ITA)

CONTACTS AND LOCATIONS:
Overall Officials: Cinzia Ferraris, PhD, Principal Investigator — University of Pavia
Locations (1):
- University of Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mills S, Brown H, Wrieden W, White M, Adams J. Frequency of eating home cooked meals and potential benefits for diet and health: cross-sectional analysis of a population-based cohort study. Int J Behav Nutr Phys Act. 2017 Aug 17;14(1):109. doi: 10.1186/s12966-017-0567-y. PMID 28818089
- [Background] Teixeira AR, Bicalho D, Slater B, Lima TM. Systematic review of instruments for assessing culinary skills in adults: What is the quality of their psychometric properties? PLoS One. 2021 Aug 9;16(8):e0235182. doi: 10.1371/journal.pone.0235182. eCollection 2021. PMID 34370729
- [Background] Teixeira AR, Camanho JSP, Miguel FDS, Mega HC, Slater B. Instrument for measuring home cooking skills in primary health care. Rev Saude Publica. 2022 Aug 29;56:78. doi: 10.11606/s1518-8787.2022056003473. eCollection 2022. PMID 36043656
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- See also: site of Laboratory of Food education — https://spmsf.dip.unipv.it/it/ricerca/laboratori-e-strumentazione/laboratorio-di-educazione-alimentare-e-nutrizione-sportiva